CLINICAL TRIAL: NCT01315275
Title: An Open-label, Multicenter, Phase IV Study of the Efficacy and Safety of Ranibizumab 0.5mg in Diabetic Patients Presenting a Visual Impairment Due to Macular Edema in Current Medical Practice
Brief Title: A Clinical Study in Current Medical Practice of the Efficacy and Safety of Ranibizumab 0.5mg in Diabetic Patients Presenting a Visual Impairment Due to Macular Edema
Acronym: LUDIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002DFR08; 2010-023315-34 (EudraCT Number)
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Visual Impairment; Macular Edema
Keywords: visual impairment; macular edema; ranibizumab; visual impairment due to macular edema
MeSH Terms: conditions — Vision Disorders; Macular Edema | interventions — Ranibizumab

ARMS (1):
- Ranibizumab (Experimental)
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab

SUMMARY:
The purpose of this study is to evaluate the proportion of patients with a 10 letters gain on Best Corrected Visual Acuity (BCVA) at 6 months in current medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >18 years of age who have signed an informed consent
* Patients with Type 1 or Type 2 diabetes mellitus (according to ADA or WHO guidelines) with HbA1c not more than 10.0% at screening (Visit 1). Patients should be on diet, exercise, and/or pharmacological treatment for diabetes.
* Patients with visual impairment due to focal or diffuse DME in at least one eye
* Central Retinal thickness on OCT ≥ 250 microns in the central subfield
* BCVA score between 78 and 39 letters, inclusively, using ETDRS-like visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160)
* Decrease in vision is due to DME and not due to other causes, in the opinion of the investigator
* Medication for the management of diabetes must have been stable within 3 months prior to randomization and is expected to remain stable during the course of the study.

Exclusion Criteria:

Ocular concomitant conditions/ diseases

* Concomitant conditions in the study eye which could, in the opinion of the investigator, prevent the improvement of visual acuity on study treatment
* Active intraocular inflammation (grade trace or above) in either eye
* Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye
* History of uveitis in either eye Systemic conditions or treatments
* Active systemic infection
* History of stroke < 3 months
* Renal failure requiring dialysis or renal transplant OR renal insufficiency with creatinine levels > 2.0 mg/dl
* Untreated diabetes mellitus
* Blood pressure systolic > 160 mmHg and diastolic > 100 mmHg
* Untreated hypertension
* Known hypersensitivity to ranibizumab or any component of the ranibizumab formulation Others
* Women of childbearing potential not using the contraception method(s) specified in this study (specify), as well as women who are breastfeeding

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2011-02; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a 10 letters gain on Best Corrected Visual Acuity (BCVA) | 6 months

SECONDARY OUTCOMES:
mean average change in BCVA from baseline | 6 months
if the letters gain after 2 injections is predictive from the letters gain at 6 months | 6 months
mean number of injections needed to obtain a 10 letters gain | 6 months
mean number of injections needed to obtain a stable visual acuity for three consecutive monthly assessments | 6 months
efficacy of ranibizumab IVT on Central Retinal Thickness (OCT) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (34):
- France (34):
  - Novartis Investigative Site, Paris, France
  - Novartis Investigative Site, Amiens
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Cesson-Sévigné
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Mantes La Joile
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Melun
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Osny
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Puilboreau
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Brieuc
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Saitnt Herblain
  - Novartis Investigative Site, St.-Jean
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
  - Novartis Investigative Site, Vannes

REFERENCES:
- See also: Journal Article for CRFB002DFR08 — http://iovs.arvojournals.org/article.aspx?articleid=2147075